CLINICAL TRIAL: NCT05285176
Title: Patients' Experiences During Endodontic Treatments Performed by Hospital Externs at the CHRU of Brest : a Qualitative Study
Brief Title: Patients' Experiences During Endodontic Treatments Performed by Hospital Externs at the CHRU of Brest
Acronym: ENDOVECU
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: ENDOVECU (29BRC21.0322)
Record Dates: First submitted 2022-03-01; First posted 2022-03-17 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Endodontic Disease
Keywords: patient; experience; stress; satisfaction; confidence
MeSH Terms: conditions — Dental Pulp Diseases; Personal Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Root canal treatment (RCT) consists in eliminating infected and / or inflammatory tissues inside the root canal system of the tooth by a chemo-mechanical preparation and then filling the latter in a three-dimensional, bacteriostatic and durable way to allow healing. This treatment is commonly carried out and can sometimes be long and tedious, as for example on molars with several roots.

According to numerous studies, patients consider endodontic treatments as one of the most stress-inducing dental procedures. Another study also reports satisfaction during root canal treatment in public health service. There is a paucity in literature about patients'experience of endodontic treatment when they are carried out by dental students.

The main objective of this study is to investigate patients' experience of root canal treatment in Brest dental university hospital through a qualitative methodology, with individual interviews, a verbatim transcription, followed by a qualitative analysis . This type of research can enable to keep a broad approach of patients' experience and to stay faithful to it.

DETAILED DESCRIPTION:
Volunteer patients are recruited during their endodontic treatment in Brest Dental Hospital. At the end of the treatment, the patients are asked to take part in an individual interview. The interview is carried out by a single investigator with the help of a question route, until data saturation. The interviews are transcribed verbatim and anonymously by the main investigator. The interviews are read by qualitative Analysis by two investigators in order to determine codes, gathered in categories. Then, the results will be written and discussed in an article.

ELIGIBILITY:
Inclusion Criteria:

* Patients of legal age who volunteered to participate in the study, having formulated their non-opposition
* Patients having been treated in the dental department of Brest dental university hospital by a dental student for an endodontic (=root canal) treatment

Exclusion Criteria:

* patient who has formulated his opposition
* patients not requiring endodontic treatment
* minor patients
* patients treated by the consultants or residents
* patients taking opioids, powerful psychotropic drugs or having taken Atarax® before the treatment or interview
* patients who are cognitively impaired or have a disability that impairs comprehension (hearing, speech)
* patients under the influence of drugs or alcohol

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Volunteer patients of Brest Dental University Hospital treated by endodontic (root canal) treatment
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2024-03-09 (Actual)

PRIMARY OUTCOMES:
Patients' experience of root canal treatment in Brest dental University hospital | day 1
  Individualized semi-directed interview, analyzed by content analysis

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Chevalier, Dr, Principal Investigator — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France

REFERENCES:
- [Background] Melgaco-Costa JL, Martins RC, Ferreira EF, Sobrinho AP. Patients' Perceptions of Endodontic Treatment as Part of Public Health Services: A Qualitative Study. Int J Environ Res Public Health. 2016 Apr 27;13(5):450. doi: 10.3390/ijerph13050450. PMID 27128932
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27128932/